CLINICAL TRIAL: NCT07190937
Title: Evaluation of Head and Neck Flexion Angle While Using a Smartphone
Brief Title: Evaluation of the Angle of Head and Neck Flexion Forward During Mobile Phone Use
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, MSc, Assistant Professor, Kutahya Health Sciences University
Other Study IDs: 2024/11-06
Record Dates: First submitted 2025-09-15; First posted 2025-09-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: kinovea; posture; smartphone use; cervical flexion angle; head flexion angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- individuals: Individuals between the ages of 18-30 who have used a smartphone for at least 1 year

SUMMARY:
The aim of this study is to investigate the effect of smartphone use on head and neck flexion angle during sitting and standing positions.

DETAILED DESCRIPTION:
With the increasing duration of smartphone use, concerns about musculoskeletal problems related to intensive use have also increased. Studies have shown that smartphone users tend to report pain symptoms in the neck and shoulder girdle, and that the severity of symptoms increases with the duration of smartphone use. Smartphone users are exposed to prolonged head and neck flexion during activities such as watching videos and texting. Maintaining this static posture for extended periods of time results in changes in cervical flexion angles. Numerous studies in the literature have found that neck and head flexion angles increase with smartphone use, and these angles increase with the duration of smartphone use. Studies in the literature have reported that head flexion angles typically range from 33 to 45 degrees during smartphone use. Smartphones, with their smaller screens, cause greater flexion angles in the cervical region compared to computer and tablet use. Therefore, it is important to assess head and neck flexion angles during smartphone use. Based on these assessments, it should be recommended that individuals choose appropriate positions. The study will include 30 individuals between the ages of 18 and 30, who use smartphones for more than one hour per day and for at least one year, and who have no physical disabilities. Before data collection begins, each participant who agrees to participate will sign a voluntary consent form. After inquiring about their demographic characteristics, smartphone usage duration, and medical history, each participant will watch a video using a designated smartphone in a laboratory setting, while their head and neck flexion angle will be measured using Kinovea Software. A 6.67-inch Xiaomi Mi 10T Pro smartphone will be used to watch the videos. The video will be a 5-minute video on water consumption (https://www.youtube.com/watch?v=nqZ0b6X_6Vs), and the participants' entire video will be recorded. The video will be watched in two different postures: standing and sitting in a backless chair. To minimize the effects of fatigue, participants will be given a 5-minute rest period between the two postures. Assessments will be conducted first while sitting and then while standing. Reference points (right lateral canthus, right tragus, C7 spinous process) will be marked with an anti-allergic erasable board marker to determine head and neck flexion angles. The angle between the line between the tragus and C7 spinous process and the vertical line passing through the C7 spinous process will be determined as the neck flexion angle. The angle between the line between the canthus and tragus and the vertical line passing through the tragus will be determined as the head flexion angle. The camera will be placed on a tripod 80 cm away from the participant, perpendicular to the sagittal plane of the participant, at a height corresponding to the level of the C7 spinous process. Participants will be instructed not to make any upper extremity movements while sitting. While standing, participants will be instructed not to reveal any movement in their lower extremities. Participants will be instructed to hold the smartphone with both hands during both postures. Before starting the study, a pilot study with five participants will be conducted to validate and calibrate the procedure. The changes in head and neck flexion angles for each participant between seconds 0, 150, and 300, and the average head and neck angle over the 5-minute period will be calculated using Kinovea Software.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 30
* Using a smartphone for more than one hour per day

Exclusion Criteria:

* Having a musculoskeletal, neurological, or mental disorder
* Having had trauma or surgery in the neck, upper, or lower extremities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Kutahya Health Sciences University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation students
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Kinovea Software | Baseline (First assessment)
  Calculation of head and neck flexion angle using Kinovea Software

CONTACTS AND LOCATIONS:
Overall Officials: Zeynel TEPE, Research Assistant, Principal Investigator — Kütahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No